CLINICAL TRIAL: NCT02125539
Title: Navigating My Journey (NmJ): A Relapse Prevention Program for Adolescents -- Field Trial
Brief Title: Field Trial of a Relapse Prevention Program for Adolescents Receiving Substance Use Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMJ 2R44DA026645-02A1; 2R44DA026645-02A1 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-04-29 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Substance-Related Disorders
Keywords: Online adolescent substance abuse relapse prevention program
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Navigating my Journey program (Experimental): Client participants of counselors who were randomized to the experimental condition will receive the following intervention: The online Navigating my Journey relapse prevention program is an adjunct to outpatient treatment. We will ask client participants to complete at least 12 Navigating my Journey sessions and discuss them with their counselors.
  Interventions: Behavioral: Navigating my Journey program
- Attention Control (Active Comparator): Client participants of counselors who were randomized to the control condition will receive their typical course of counseling and a link to online online health information in PDF form as an attention control.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Navigating my Journey program — The online relapse prevention program called Navigating my Journey is designed for adolescents who are receiving outpatient treatment for substance abuse. Since the Navigating my Journey program will be available to adolescents 24/7, it is easy for them to access at their convenience. The program functions as an adjunct to treatment and is designed to complement and enhance the work the adolescent does with the counselor during counseling sessions. The core intervention is expected to last for 12 weeks.
  Arms: Navigating my Journey program
Behavioral: Attention Control — Client participants in the control group will receive their typical course of counseling and a link to online online health information in PDF form as an attention control.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to provide a comprehensive evaluation of the new, Navigating my Journey program for adolescents receiving treatment in an outpatient substance abuse center.

The primary hypotheses are that, relative to the control condition, Navigating my Journey will be associated with significantly higher motivation, higher self-efficacy, improved relapse coping skills, and lower substance use. The secondary hypotheses are that, relative to the control condition, Navigating my Journey will be associated with increased therapeutic alliances with counselors.

DETAILED DESCRIPTION:
The randomized, control trial will compare clients receiving treatment in an outpatient substance abuse center in the following two conditions -- (1) Experimental: Navigating my Journey (includes 12 core lessons and 8 supplemental lessons); and (2) Attention Control (treatment as usual plus online health information) -- using a longitudinal design.

ELIGIBILITY:
Inclusion Criteria:

* currently meeting with a counselor in the study at least twice per month during the next 3 months
* age 13 to 21
* ability to read and speak English
* have drugs and/or alcohol as their primary or secondary substance used
* have completed detox as necessary
* an active email account.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Substance Use Across Time | Baseline, 1 month post baseline, 3 months post baseline, 6 months post baseline
  Participants will be asked how many days in the past 30 days they used a variety of substances, including alcohol. This self report question format is widely used to assess substance use (e.g., the GPRA from CSAT; SAMHSA, 2010).
Change in Motivation to Change Across Time | Baseline, 1 month post baseline, 3 months post baseline, 6 months post baseline
  The 32-item University of Rhode Island Change Assessment Questionnaire (URICA; McConnaughy et al., 1983, 1989) will be used to measure motivation to change. It has four 8-item scales (Precontemplation, Contemplation, Action, and Maintenance) that can be combined to create a single Readiness to Change score (C + A + M - PC = Readiness). Participants rate each item 1=Strongly Disagree to 5=Strongly Agree. This scale has good reliability and validity with adolescents (Greenstein et al., 1999).
Change in Self-Efficacy Across Time | Baseline, 1 month post baseline, 3 months post baseline, 6 months post baseline
  Drug Avoidance Self-Efficacy Scale (DASES). The DASES (Martin et al., 1995) assesses one's current self-efficacy to resist drug use in hypothetical high-risk situations. The scale contains 16 items, and responses are rated on a 7-point scale ranging from "certainly yes" to "certainly no."
Change on the Adolescent Relapse Coping Questionnaire (ARCQ) Across Time | Baseline, 1 month post baseline, 3 months post baseline, 6 months post baseline
  The ARCQ (Myers et al., 2006) assesses "temptation coping responses among adolescents." It begins with a short assessment of appraisal (5 items total) of a situation where peers are drinking and using, followed by 28 items rated between 1 = Definitely would not do or think, through 7 = Definitely would do or think. These 28 items comprise three subscales: Cognitive and behavioral problem solving (e.g., Let your feelings out somehow; alpha = .82); Self-critical thinking (e.g., Criticize or lecture yourself; alpha = .80); and Abstinence-focused coping (e.g., Leave or avoid the situation; alpha = .78).

SECONDARY OUTCOMES:
Change in Therapeutic Alliance Across Time | Baseline, 1 month post baseline, 3 months post baseline, 6 months post baseline
  Working Alliance Inventory-Short Form (Clients) (WAI-S). The working alliance between counselor and client is a critical indicator of client outcomes. The WAI-S (Tracey & Kokotovic, 1989) is a short form (12 items) of the original WAI (36 items). It has three sub-scales - therapeutic bond, agreement on tasks, and agreement about goals. Items are scored on a 7-point scale (1 = rarely to 7 = always, range 12-84).
Client Satisfaction | 3 months post baseline
  At the end of the study, participants will be asked to evaluate the resources they reviewed (i.e., attention control materials or Navigating my Journey program) and their experience in the study. Because this survey is dependent on content and features which will have been developed in Phase II, it will be fully developed at that time. We expect that participants will rate the program's usability (ease of navigation, information organization, and graphical interface) and content (relevance, interest, comprehension) on a 5-point Likert scale (1 = not at all to 5 = extremely). Examples of questions that may be included are: To what degree were these resources helpful in your treatment? How helpful were these resources in preparing you to deal with the challenges you face in recovery? How helpful these resources in keeping you involved in treatment?
Change in Client Engagement/Attendance Across time | 1 month post baseline and 6 months post baseline
  Counselors will be asked to fill out a form to indicate if the client is still in treatment at the center and if so, how many sessions each participant attended since the last status update. If the client is no longer receiving treatment at the center, we will ask why the participant is not still in treatment at the center and if there were any other factors affecting their discharge. Each form is expected to take less than 10 minutes.
Counselor Satisfaction | 3 months post baseline
  At the end of the study, counselors will be asked to evaluate the resources they viewed and their experience in the study via an online questionnaire and phone interview. These activities will take a maximum of 60 minutes. Participants will rate (1) the degree to which these resources helped to make improvements in their clients' outcomes; (3) the effectiveness of these resources in dealing with the challenges of recovery; (4) overall, what they thought of these resources; (5) the ability of these resources to engage their substance abuse clients; (6) how likely they are to recommend these resources to a colleague; and (7) what improvements they would recommend to make these resources better to help in substance abuse treatment. Feedback from counselors in the experimental condition will be used to make modifications to Navigating my Journey before marketing occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberlee Trudeau, Ph. D., Principal Investigator — Inflexxion, Inc.
Locations (1):
- Inflexxion, Inc., Newton, Massachusetts, United States